CLINICAL TRIAL: NCT05941702
Title: Feasibility and Acceptability of Body Signal Integration Training for Functional Neurological Disorder: A Case Series
Brief Title: Body Signal Integration Training: A Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Krishna Panchmatia, Trainee Clinical Psychologist, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KPanchmatia
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Functional Neurological Disorder
Keywords: Intervention; Interoception; Body Awareness
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Intervention Model Description: Case Series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Full session plan of the 8 sessions is uploaded to documents. This arm will consist of weekly 1 hour 1:1 sessions with Trainee Clinical Psychologist doing exercises aimed at improving interoception. Exercises will include tuning into the body under different circumstances e.g., while having a drink, looking at pictures to induce a positive mood state.
  Interventions: Behavioral: Body Signal Integration Training

INTERVENTIONS:
Behavioral: Body Signal Integration Training — Information and protocol uploaded to documents.

SUMMARY:
The goal of this clinical trial is to learn about an intervention package in individuals with Functional Neurological Disorder (FND). The main questions it aims to answer are:

* Is the intervention package acceptable to and feasible to deliver to individuals with FND?
* Does the intervention package improve symptoms of FND?

Participants will be asked to engage in 8 weekly sessions of an intervention aimed to improve the perception of signals coming from the body (interoception). Participants will be asked to complete tasks between session practising tuning into signals from the body. Participants will also be asked to complete questionnaires measuring their psychological wellbeing, FND symptoms and interoception.

DETAILED DESCRIPTION:
The designed intervention is derived from the Integrative Cognitive Model (ICM) of medically unexplained symptoms and Psychogenic Non-Epileptic Seizures, (Brown, 2004; Ven den Bergh, Witthoft, Petersen, & Brown, 2017; Brown & Reuber, 2016). This model suggests that conscious body perceptions are interpretations of bottom-up signals influenced by top-down factors such as attention, beliefs, fears and emotional states. The model suggests that Functional Neurological Disorders are distortions in body awareness that arise when normal bodily signals are misinterpreted as noxious, due to a combination of top-down factors and the bodily signals themselves being weak. The proposed intervention targets several factors identified as important in this model, including imprecise bodily signals, poor emotion recognition and regulation, anxious beliefs and fears about symptoms and symptom-focussed processing. The intervention aims to sharpen signals from the body by reducing avoidance and misinterpretation of those signals and thereby improve body perception and interoceptive accuracy. If acceptable, feasible and effective, the proposed intervention would contribute to the literature for the Integrative Cognitive Model of FND and inform future interventions for individuals with FND.

Participants will be offered 8, 1-hour, online sessions, delivered weekly via Microsoft Teams. The psychological intervention will focus on developing skills to improve attunement to the signals from the body to the brain.

* The sessions will involve engaging in various exercises tuning into the body under different circumstances. Participants will be asked to tune into how particular objects feel in their hands. Participants may be presented with images or scenarios to make them feel a little happy or sad and then will be asked to tune into how the body feels in response to them.
* Participants will be asked to complete weekly measures online via Qualtrics survey, they will be asked to do this in the 10-15 minutes prior to their session commencing.
* A full manual of the intervention plan will be uploaded to documents.
* Following the final session of treatment, a date to complete a one-month follow up will be arranged with the participant.

Follow-Up:

* One month following the end of psychological therapy, a session will be attended remotely via Microsoft Teams by participants.
* During this session, all pre-treatment, weekly and post-treatment measures will be re-administered including questionnaires measuring satisfaction with therapy.

ELIGIBILITY:
Inclusion Criteria:

* Currently experiencing FND symptoms, as measured on items 34-47 on the SOMS-7 (excluding seizures and hallucinations). The study is aiming to investigate the feasibility of an intervention for individuals with FND.
* Confirmation of diagnosis of FND (through letter from medical doctor) to ensure participants have a diagnosis of FND and are therefore the target audience for the intervention
* Willing and able to participate in remote therapy. The intervention will be delivered remotely so participants must be willing to engage with remote therapy.
* Able to converse in English proficiently without support from a link worker. The study will not be using interpreters and so an ability to converse proficiently in English to be able to engage with the intervention is needed.
* Residing in the UK for the duration of the study, this is in order to develop crisis and risk management plans for participants should they experience any negative effects from therapy or any risks be expressed throughout the course of the intervention.

Exclusion Criteria:

* Currently undergoing any other psychological therapy
* Previous experience of a mindfulness-based intervention targeting FND.
* Individuals with symptoms of epilepsy and loss of consciousness.
* Symptoms of psychosis (as assessed on the Comprehensive Assessment of At-Risk Mental State, CAARMS).
* Diagnosis of any type of Personality Disorder
* Active plans of self-harm and/or suicide. Potential participants will be asked to complete the risk items on the CORE-OM and will be interviewed around these. This is to ensure the safety of participants engaging in novel therapy and to manage the risks of any potential adverse side-effects of therapy
* History of prior suicide attempts, to manage the risks of causing negative side effects of therapy
* Any difficulties with alcohol or substance misuse.
* Individuals with active symptoms of Post Traumatic Stress Disorder (PTSD) i.e., having current symptoms of nightmares and flashbacks.
* Individuals with symptoms of an eating disorder.

Rationale for exclusion criteria is described in the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Panchmatia, Principal Investigator — University of Manchester
Locations (1):
- Krishna Panchmatia, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 8
Completed | 7 (Completion of all treatment sessions (8 sessions, weekly))
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 4
  Caribbean | 1
  Black/Black British/Caribbean | 1
  Mixed Ethnicity | 1
  White European | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Complete 80% of the Intervention
Description: This is a measure of adherence to the intervention. 80% of participants attending 80% of sessions offered will be considered acceptable adherence
Time Frame: 8 weeks (span of intervention delivery)
Population: Number of participants that completed intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 8
Participants | 7

2. Primary Outcome: Number of Participants Rating the Therapy as Acceptable on Questionnaire of Therapy Satisfaction
Description: Measure of acceptability of intervention
Time Frame: 8 weeks (span of intervention delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 7
Participants | 7

3. Primary Outcome: Number of Serious Adverse Reactions as Evidenced by Significant Increase in Distress or Symptom Rating on Euroqol Health Questionnaire (EQ5D), Clinical Outcomes in Routine Evaluation (CORE-10) or FND Questionnaire
Description: Number of serious adverse reactions will be a measure of feasibility and acceptability of the intervention
Time Frame: 8 weeks (span of the intervention delivery)
Population: Number of participants that experienced adverse reaction to treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 8
Participants | 0

4. Secondary Outcome: Number of Participants Showing a Reliable Change Reduction in Core FND Symptoms as Measured by Screening for Somatic Symptom Disorders (SOMS-7)
Description: Measure of treatment efficacy
Time Frame: Approximately 3 months - measure will be from baseline measure completion to end of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 7
Participants | 3

5. Secondary Outcome: Number of Particip
Description: Number of Participants with a Clinically Significant Change of Interoception Measuring Treatment Efficacy
Time Frame: Approximately 3 months - measure will be from baseline completion until end of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 7
Participants | 5

ADVERSE EVENTS:
Time Frame: 3 months
Description: No unanticipated adverse events occurred or serious adverse events occurred. One individual reported increased awareness of FND symptoms and associated distress, they chose to drop out of the study and subsequently contacted researchers to inform symptoms had resolved - this was deemed an 'anticipated adverse reaction' to treatment. No further events/reactions occurred during the trial
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=8)
Psychological Distress (Social circumstances) | 1 (1) — Stress caused by tuning into the body leading to greater perception of symptoms/distress associated with symptoms. In this instance,

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT05941702/Prot_SAP_002.pdf
  • Informed Consent Form (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT05941702/ICF_001.pdf